CLINICAL TRIAL: NCT01579110
Title: Efficacy and Safety of Levamisole Combined With Standard Prednisolone in Warm Antibody Autoimmune Hemolytic Anemia.
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Institute of Hematology & Blood Diseases Hospital, China (Other)
Responsible Party: Principal Investigator, Yizhou Zheng, Vice director of the therapeutic centre of anemic diseases, Institute of Hematology & Blood Diseases Hospital, China
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ZXMZ2012
Record Dates: First submitted 2012-04-13; First posted 2012-04-17 (Estimated); Last update posted 2012-04-19 (Estimated); Status verified 2012-04

CONDITIONS: Anemia; Anemia, Hemolytic; Anemia, Hemolytic, Autoimmune; Hemolysis; Hematologic Diseases; Autoimmune Diseases; Immune System Diseases; Pathologic Processes
Keywords: autoimmune hemolytic anemia; hemolytic anemia; Levamisole; Treatment of autoimmune hemolytic anemia; warm antibody dependant autoimmune hemolytic anemia
MeSH Terms: conditions — Anemia; Anemia, Hemolytic; Anemia, Hemolytic, Autoimmune; Hemolysis; Hematologic Diseases; Autoimmune Diseases; Immune System Diseases; Pathologic Processes | interventions — Levamisole; Prednisone

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- prednisolone + levamisole (Experimental)
  Interventions: Drug: levamisole
- Prednisone (Active Comparator)
  Interventions: Drug: Prednisone

INTERVENTIONS:
Drug: levamisole — Levamisole 2.5mg/kg(every other day) over six months.
  Prednisone 1mg/kg for two weeks and then tapered off dosage over two months.
  Arms: prednisolone + levamisole
Drug: Prednisone — Prednisone 1mg/kg for two weeks and then tapered off dosage over two months.
  Arms: Prednisone

SUMMARY:
The purpose of this study is to determine whether Levamisole plus prednisone can further improve the efficacy，extend the remission duration and reduce the dosage of prednisone for newly diagnosed warm antibody autoimmune hemolytic anemia.

DETAILED DESCRIPTION:
The first line treatment in warm antibody autoimmune hemolytic anemia (WAIHA) is the glucocorticoid, but most of the patients, hemolytic events will frequently recurred after end of treatment or during the gradual reduction in dosage of prednisolone. As a result, many patients will finally accepted long-term glucocorticoids or other immunosuppressive drugs. How to reduce the relapse rate of AIHA is still difficult. Levamisole（LMS）is a immunoregulator.Recent studies have shown LMS has been widely used to treat autoimmune diseases ,such as rheumatoid arthritis, systemic lupus erythematosus and idiopathic thrombocytopenic purpura. The purpose of this study is to determine whether LMS combined with prednisolone can further improve the efficacy，extend the remission duration and reduce the dosage of prednisone for newly diagnosed warm antibody autoimmune hemolytic anemia.

ELIGIBILITY:
Inclusion Criteria:

* Clinical and biochemical signs of hemolytic anaemia
* Positive Coombs test with anti-IgG or and with anti-CD3d
* Newly diagnosed Warm Autoimmune Hemolytic Anemia
* Adequate contraceptive measures for women of childbearing potential
* informed consent signed

Exclusion Criteria:

* Active infection which requires antibiotic treatment
* Pregnant or lactating women
* Epilepsy and mental illness
* Kidney and liver function abnormal

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2012-04; Primary Completion 2015-04 (Estimated); Study Completion 2016-04 (Estimated)

PRIMARY OUTCOMES:
Number of patients in each group in complete or partial remission | one year

SECONDARY OUTCOMES:
Side effects | 1year

CONTACTS AND LOCATIONS:
Overall Officials: Yizhou Zheng, doctor, Principal Investigator — Blood Diseases Hospital Chinese Academy of Medical Sciences
Locations (1):
- Blood Diseases Hospital Chinese Academy of Medical Sciences, Tianjin, Tianjin Municipality, China